CLINICAL TRIAL: NCT01359189
Title: Initial Exploratory Evaluation of a Transrectal Scintigraphic Detector (ProxiScanTM) for Detection of Primary Prostate Cancer Utilizing a Prostate Specific Membrane Antigen (PSMA) Based Radiotracer (ProstaScint®)
Brief Title: Evaluation of a Transrectal Scintigraphic Detector(ProxiScanTM) for Detection of Primary Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J1050
Record Dates: First submitted 2011-05-19; First posted 2011-05-24 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Suspected Primary Prostate Cancer
Keywords: Suspected Primary Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Suspected Primary Prostate Cancer (Experimental): Patients with suspected prostate cancer will be evaluated for initial proof of concept and feasibility of a scintigraphic rectal probe (ProxiScanTM) utilizing a PSMA receptor radiopharmaceutical (ProstaScint®). To explore the adjunctive benefit/feasibility of PSMA distribution in the normal prostate versus prostate cancer gland utilizing TRUS and CT/SPECT hybrid imaging, biopsy negative patients will be considered as normal controls. This is an exploratory, open label trial and randomization is not required. Subject blinding is not needed and investigator blinding in not possible.
  Interventions: Device: ProxiScan (scintigraphic rectal probe)

INTERVENTIONS:
Device: ProxiScan (scintigraphic rectal probe) — ProxiScanTM is a compact, high-resolution gamma camera which has been developed for the detection of cancer and other abnormalities in the body by imaging the distribution of radionuclides in the human body using planar imaging techniques. This camera is capable of high-performance imaging of radiopharmaceuticals distributed within anatomical regions of interest located close to the camera head. The ProxiScan compact scintigraphic detector was approved by the FDA to market the device for the following indication: "The ProxiScanTM is indicated for use in imaging the distribution of radionuclides in the human body using planar imaging techniques. ProxiScanTM may also be used intraoperatively, on pathological specimens and for endocavity applications if a protective sheath is used."

SUMMARY:
This is a feasibility, exploratory, and proof-of-concept study to evaluate rectal probe scintigraphy device (ProxiScanTM) to detect PSMA specific radiopharmaceutical agent (ProstaScint®) in patients with suspected primary prostate cancer. ProxiScanTM is a small cadmium zinc telluride (CST)-based compact gamma camera the size of a trans-rectal ultrasound (TRUS) developed by Hybridyne Imaging Technologies, Inc.To explore the adjunctive benefit/feasibility of PSMA distribution in the normal prostate versus prostate cancer gland utilizing TRUS and CT/SPECT hybrid imaging, biopsy negative patients will be considered as normal controls. Prostate cancer sextant biopsy histology results will be correlated with ProxiScanTM, TRUS, and pelvis planar and SPECT/CT. Our hypothesis is that it will be safe and feasible to utilize a rectal probe scintigraphy (ProxiScanTM) to detect PSMA specific ProstaScint® uptake in primary prostate cancer.

DETAILED DESCRIPTION:
This is a feasibility, exploratory, and proof-of-concept study to evaluate rectal probe scintigraphy device (ProxiScanTM) to detect PSMA specific radiopharmaceutical agent (ProstaScint®) in patients with suspected primary prostate cancer. ProxiScanTM is a small cadmium zinc telluride (CST)-based compact gamma camera the size of a trans-rectal ultrasound (TRUS) developed by Hybridyne Imaging Technologies, Inc. Due to its inherent small size, this camera is capable of potentially imaging of prostate cancer specific radiopharmaceutical uptake distributed within the prostate gland located closely adjacent to the camera head.In this study the investigators will enroll patients with a clinical suspicion and high likelihood of prostate cancer. A scintigraphic rectal probe (ProxiScanTM) will be used to detect ProstaScint® uptake in the prostate gland, in comparison to TRUS and pelvis planar and SPECT/CT. The incidence of biopsy positive prostate cancer in patients with suspected disease clinically can range from 25% to 40%; therefore up to 12 patients will be enrolled on this study. To explore the adjunctive benefit/feasibility of PSMA distribution in the normal prostate versus prostate cancer gland utilizing TRUS and CT/SPECT hybrid imaging, biopsy negative patients will be considered as normal controls. Prostate cancer sextant biopsy histology results will be correlated with ProxiScanTM, TRUS, and pelvis planar and SPECT/CT. Our hypothesis is that it will be safe and feasible to utilize a rectal probe scintigraphy (ProxiScanTM) to detect PSMA specific ProstaScint® uptake in primary prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Elevated PSA ≥ 4ng/mL and/or abnormal digital rectal exam suspicious for prostate cancer.
* Planned sextant prostate biopsy.
* Sufficient time period to complete the imaging protocol and 5 to 7 day safety follow-up assessment without prostate biopsy or therapeutic intervention.
* Patient is judged by the Investigator to have the initiative and means to provide written consent and be compliant with the protocol and be able and commits to make the required study visits.
* Ambulatory with ECOG performance status of 0 or 1; or Karnofsky performance scale of ≥ 70. (seen appendix below)
* Patient is between 30 and 75 years of age.

Exclusion Criteria:

* Patient or physician plans definitive concomitant chemotherapy, therapeutic radiation treatment, biologic treatment and/or local ablative treatment for cancer within the interval of study participation.
* Prior therapeutic pelvic irradiation.
* Recent prostate biopsy, within 1 month of study enrollment.
* Patient with contraindications to TRUS-guided prostate biopsy (continuous need for anti-coagulation, no rectum, etc.)
* Clinical evidence of prostatitis, or other benign prostate gland abnormality, that would explain elevated PSA and/or (digital rectal exam) DRE findings.
* Active malignancy or therapy for malignancy within 6 months, other than basal or squamous cell carcinoma of the skin.
* Patient received a radiopharmaceutical which was within 5 physical half-lives at the time of study imaging.
* Known history of human-anti-murine-antibodies (HAMA) or known allergic reaction to previously received murine based products.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of a Transrectal Scintigraphic Detector (ProxiScanTM) to detect and localize prostate specific membrane antigen (ProstaScint®) radiotracer uptake in suspected primary prostate cancer patients. | 12 months
  The proximity of the placement of the ProxiScanTM device to the prostate should result in an improvement in the sensitivity and specificity for detection of prostate cancer specific radiopharmaceutical detection. The primary objectives will be evaluated at the patient level, while secondary objectives will be analyzed based on data and outcomes measured by region of the prostate (sextant).

SECONDARY OUTCOMES:
TRUS, ProxiScan and SPECT/CT when compared to biopsy | 12 months
  Secondary Objectives:
  1. Estimate the sensitivity and specificity for three methods of detection: TRUS, ProxiScan and SPECT/CT when compared to biopsy.
  2. Estimate the sensitivity and specificity for ProxiScan and SPECT/CT when compared to PSMA IHC measurements.
  3. If prostatectomy histology results are available, the ability to detect areas of cancer among multiple slices of prostate tissue with TRUS, SPECT/CT and ProxiScan will be evaluated.
  4. Explore reclassification properties of the ProxiScan results compared to the SPECT/CT at the patient level.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Cho, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States